CLINICAL TRIAL: NCT03685019
Title: Optimum Radiographic Assessment of the Medial and Lateral Tibiofemoral Compartments Within the Arthritic Knee
Brief Title: Optimum Radiographic Assessment of the Knee
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Thomas Hamilton, Primary investigator, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 256
Record Dates: First submitted 2015-05-07; First posted 2018-09-26 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Each of the interventions was planned to be applied in sequence.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Valgus stress - lateral compartment (Experimental): Valgus stress radiograph. Joint space width measured in lateral compartment.
  Interventions: Radiation: Valgus Stress
- Varus stress - medial compartment (Experimental): Varus stress radiograph. Joint space width measured in medial compartment.
  Interventions: Radiation: Varus stress
- 0 degree flexion - medial compartment (Experimental): 0 degree flexion radiograph. Joint space width measured in medial compartment.
  Interventions: Radiation: 0 degree flexion radiograph
- 0 degree flexion - lateral compartment (Experimental): 0 degree flexion radiograph. Joint space width measured in medial compartment.
  Interventions: Radiation: 0 degree flexion radiograph
- 20 degree flexion - medial compartment (Experimental): 20 degree flexion radiograph. Joint space width measured in medial compartment.
  Interventions: Radiation: 20 degree flexion radiograph
- 20 degree flexion - lateral compartment (Experimental): 20 degree flexion radiograph. Joint space width measured in lateral compartment.
  Interventions: Radiation: 20 degree flexion radiograph
- 45 degree flexion - medial compartment (Experimental): 45 degree flexion radiograph. Joint space width measured in medial compartment.
  Interventions: Radiation: 45 degree flexion radiograph
- 45 degree flexion - lateral compartment (Experimental): 45 degree flexion radiograph. Joint space width measured in lateral compartment.
  Interventions: Radiation: 45 degree flexion radiograph

INTERVENTIONS:
Radiation: Valgus Stress — Valgus stress radiograph
  Arms: Valgus stress - lateral compartment
Radiation: Varus stress — Varus stress radiograph
  Arms: Varus stress - medial compartment
Radiation: 0 degree flexion radiograph — 0 degree flexion radiograph
  Arms: 0 degree flexion - lateral compartment; 0 degree flexion - medial compartment
Radiation: 20 degree flexion radiograph — 20 degree flexion radiograph
  Arms: 20 degree flexion - lateral compartment; 20 degree flexion - medial compartment
Radiation: 45 degree flexion radiograph — 45 degree flexion radiograph
  Arms: 45 degree flexion - lateral compartment; 45 degree flexion - medial compartment

SUMMARY:
X-rays are the most frequently used imaging test when evaluating the knee for joint replacement. They are non-invasive, safe and cost effective. They allow assessment of: progression of disease, appropriateness for joint replacement, in particular unicompartmental knee replacement (UKR), as well as likely prognosis following replacement. Despite a multitude of standardised views there is a lack of consensus regarding the optimum views to evaluate joint space narrowing within each compartment (lateral, medial and patellofemoral).

This study will evaluate the status of knee cartilage in 225 patients with varying degrees, and patterns, of knee osteoarthritis (OA) using standing extension anteroposterior, 15 degrees flexion posteroanterior, 45 degrees flexion posteroanterior and valgus and varus stress views as well as MRI. These results will be compared to the gold standard imaging technique of stress views as well as to direct measurements of retrieved tissue in those patients who undergo knee replacement surgery. The sensitivity and specificity of each of the imaging techniques at predicting suitability for UKR will be calculated, the optimum imaging views proposed, and ultimately the results of this study will be used to develop a decision aid, based on optimum views, to help clinicians decide between likelihood of a patient being a candidate for UKR based on pre-operative X-ray findings.

DETAILED DESCRIPTION:
The optimum imaging protocol is one that is acceptable to patients, involves the fewest X-rays to obtain the most clinically relevant information and one that utilizes the least resources in terms of staff and equipment. Currently standard assessment involves: standing anteroposterior, lateral and skyline views. In addition in patients being considered for joint replacement valgus/varus stress X-rays are used to evaluate the lateral compartment (as well as medial collateral ligament) and medial compartment respectively to assess the status of the cartilage. In patients with loss of cartilage on one side, typically medial, but preserved cartilage on the other a UKR, as opposed to total knee replacement (TKR), may be indicated.

Currently there is a lack of consensus amongst orthopaedic surgeons as to the best way to image the knee joint to establish degree and pattern of arthritis. For a long time it has been known that weight bearing views are a better method at establishing the true joint space compared to non-weight bearing views width due to the increased forces across the joint. In addition it is known that full extension views, despite being the most commonly used view, may also underestimate joint space narrowing as in full extension the femur and tibia articulate across an area of the joint that is not typically not involved during activity, and hence can have relatively well preserved cartilage, giving a false impression of the joints disease state. These findings have been adopted, and continue to be adopted, into routine clinical practice and there continues to be an increase in the proportion of surgeons performing standing and semi-flexed views. However the best method of evaluating the disease state in each compartment has yet to be defined.

When deciding between UKR and TKR the detection of the degree and pattern of arthritis is of critical importance. UKR are known to perform poorly in partial thickness disease and require full thickness cartilage in the retained tibiofemoral compartment. To establish whether a patient meets the indications for UKR X-rays are used with stress views being the gold standard, as well as the standard assessment that the studies of long term outcomes on UKR are based. Gibson and Goodfellow, who were first to describe stress X-rays in the workup of a patient for UKR, reported that those patients with a joint space width of more than 5mm in the lateral compartment had intact lateral cartilage during surgery making them appropriate for UKR. More recently Waldstein et al. reported that patients with a lateral joint space width of more than 4mm may be appropriate for UKR however overall they noted poor correlation between joint space width measured on valgus stress views and intra-operative Outerbridge grade.

In addition to the low quantity of evidence regarding the relationship between stress views and intra-operative status of the joint the feasibility of performing stress X-rays also limits their use. Stress X-rays are resource dependent, can be uncomfortable for patients and require an additional practitioner. As such they are often not performed with many clinicians adopting alternative X-ray views, MRI or direct observation via arthroscopy. It has been proposed that standing views with the knee in 15 degrees then 45 degrees flexion may load the medial and lateral compartments respectively and that these views may be an alternative to stress views without the requirement for an additional practitioner. However the outcomes based on these forms of assessment, and the relationship between the joint space width measured using these contemporary techniques has not been reported. An alternative would include a stress device that allows a stress X-ray to be performed without the requirement of the clinician.

This study will evaluate the status of knee cartilage in 225 patients with varying degrees, and patterns, of knee OA using standing extension anteroposterior, 15 degrees flexion posteroanterior, 45 degrees flexion posteroanterior and valgus and varus stress views as well as MRI. These results will be compared to the gold standard imaging technique of stress views as well as to direct measurements of retrieved tissue in those patients who undergo knee replacement surgery. The sensitivity and specificity of each of the imaging techniques at predicting suitability for UKR will be calculated, the optimum imaging views proposed, and ultimately the results of this study will be used to develop a decision aid, based on optimum views, to help clinicians decide between likelihood of a patient being a candidate for UKR based on pre-operative X-ray and MRI findings.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis any grade, affecting the tibio-femoral joint
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 50 years or above.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Previous joint replacement on ipsilateral knee
* Previous anterior cruciate ligament reconstruction or injury
* Previous high tibial osteotomy
* Previous intraarticular fracture
* History of Inflammatory arthritis
* Unable to stand with assistance for two minutes

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

REFERENCES:
- See also: Oxford Orthopaedic Engineering Centre, Nuffield Department of Orthopaedics, Rheumatology and Musculoskeletal Sciences (NDORMS), University of Oxford — https://www.ndorms.ox.ac.uk/research-groups/oxford-orthopaedic-engineering-centre

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight participants recruited with each undergoing treatment in each arm
Groups:
- All Participants: All participants undergoing:
  Valgus stress Varus stress 0 degree flexion medial compartment 0 degree flexion lateral compartment 20 degree flexion medial compartment 20 degree flexion lateral compartment 45 degree flexion medial compartment 45 degree flexion lateral compartment
Period: Valgus Stress (Lateral Compartment)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0
Period: Varus Stress (Medial Compartment)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0
Period: 0 Degrees Flexion (Medial Compartment)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0
Period: 0 Degrees Flexion (Lateral Compartment)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0
Period: 20 Degrees Flexion (Medial Compartment)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0
Period: 20 Degrees Flexion (Lateral Compartment)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0
Period: 45 Degrees Flexion (Medial Compartment)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0
Period: 45 Degrees Flexion (Lateral Compartment)
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 70 [63 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Knee Minimum Joint Space Width (Medial and Lateral Compartment)
Description: Knee minimum joint space width (medial and lateral compartment) measured using custom, validated, in house software (KneeMorph, MATLAB, MathWorks, Massachusetts).
Time Frame: Day 0
Population: Participants were recruited for the trial but due to poor recruitment and logistical challenges none of the participants underwent any of the proposed assessments and as such no outcome data was collected. The trial terminated due to poor recruitment.
Arm/Group | Valgus Stress - Lateral Compartment | Varus Stress - Medial Compartment | 0 Degree Flexion - Medial Compartment | 0 Degree Flexion - Lateral Compartment | 20 Degree Flexion - Medial Compartment | 20 Degree Flexion - Lateral Compartment | 45 Degree Flexion - Medial Compartment | 45 Degree Flexion - Lateral Compartment
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Sensitivity and Specificity of X-ray Views at Demonstrating Full Thickness Cartilage Loss, Partial Thickness Cartilage Loss and Preserved Full Thickness Cartilage Within Each Compartment (Medial & Lateral) of the Knee
Description: The gold standard will be grade of arthritis at time of surgery in those patients undergoing knee replacement as part of their routine clinical care.
  Each compartment will be graded independently. An X-ray demonstrating a joint space width (JSW) of 0mm will be classified as full thickness cartilage loss, a JSW of >0mm but <4mm will be classified as partial thickness cartilage loss and a JSW of 4mm or greater will be classified as preserved full thickness cartilage.
  The sensitivity of each view at predicting the observed grade of cartilage disease within each compartment at the time of surgery will be recorded.
Time Frame: Day 0
Population: as for outcome 1
Arm/Group | Valgus Stress - Lateral Compartment | Varus Stress - Medial Compartment | 0 Degree Flexion - Medial Compartment | 0 Degree Flexion - Lateral Compartment | 20 Degree Flexion - Medial Compartment | 20 Degree Flexion - Lateral Compartment | 45 Degree Flexion - Medial Compartment | 45 Degree Flexion - Lateral Compartment
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse event and/or serious adverse event related to positioning for imaging.
Arm/Group | Valgus Stress - Lateral Compartment | Varus Stress - Medial Compartment | 0 Degree Flexion - Medial Compartment | 0 Degree Flexion - Lateral Compartment | 20 Degree Flexion - Medial Compartment | 20 Degree Flexion - Lateral Compartment | 45 Degree Flexion - Medial Compartment | 45 Degree Flexion - Lateral Compartment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03685019/Prot_SAP_000.pdf